CLINICAL TRIAL: NCT00131352
Title: A Multi-Centre, Parallel, Double-Blind, Blinded Evaluator, Randomised, Placebo-Controlled Evaluation of the Efficacy and Safety of a Single Dose of 6 mL of Synvisc in Patients With Symptomatic Osteoarthritis of the Knee
Brief Title: A Study of the Safety and Efficacy of Hylan G-F 20 (Synvisc) in Patients With Symptomatic Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYNV00704
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis, Knee; Musculoskeletal Diseases
Keywords: Osteoarthritis of the knee; Musculoskeletal
MeSH Terms: conditions — Osteoarthritis, Knee; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synvisc (Experimental): Participants with symptomatic primary osteoarthritis (OA) of the knee received a single injection of 6 mL hylan G-F 20 (Synvisc).
  Interventions: Device: hylan G-F 20
- Saline Control (Placebo Comparator): Participants (control group) with symptomatic primary osteoarthritis (OA) of the knee received a single injection of 6 mL phosphate buffered saline.
  Interventions: Other: Phosphate Buffered Saline

INTERVENTIONS:
Device: hylan G-F 20 — Single injection of 6 mL of hylan G-F 20 (Synvisc).
  Other Names: Synvisc-One
  Arms: Synvisc
Other: Phosphate Buffered Saline — Single injection of 6 mL phosphate buffered saline.
  Arms: Saline Control

SUMMARY:
This clinical study is to evaluate the safety and efficacy of hylan G-F 20 (Synvisc) in patients with symptomatic knee osteoarthritis (OA). Patients will be given 6 mL of hylan G-F 20 (Synvisc) (or a phosphate buffered saline control), with a possible repeat treatment with Synvisc after the week 26 visit.

DETAILED DESCRIPTION:
The trial included an initial 26 week treatment with 6 mL of hylan G-F 20 (Synvisc) (or a phosphate buffered saline control) followed by a 4 week repeat treatment of Synvisc.

ELIGIBILITY:
Inclusion Criteria:

* Patient with documented diagnosis of primary osteoarthritis (OA) of the target knee made at least 3 months prior to Screening,
* Has radiographic evidence of OA in the tibio-femoral compartment of the target, knee with at least 1 definite osteophyte and a measureable joint space, as diagnosed by standard X-rays taken not longer than 3 months prior to Screening, and before any baseline assessment,
* Has continued target knee pain despite conservative treatment (e.g. weight reduction, physical therapy, analgesics),
* Has pain in the target knee as demonstrated by a score of 2 or 3 on the Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale Version 3.1 (WOMAC LK 3.1) A1 (Walking Pain) Subscale ,
* Has a mean score of 1.5 to 3.5 on the Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale Version 3.1 (WOMAC LK 3.1) A (Pain) Subscale.
* Inclusion Criteria for Repeat Phase: Must have no major safety concerns during the first course of treatment as assessed by the Investigator; Must have a WOMAC LK 3.1 A score of at least 1.

Exclusion criteria:

* Has modified Kellgren-Lawrence Numerical Grading System of grade IV in the patello-femoral compartment of the target knee confirmed by standard X-rays taken not longer than 3 months prior to Screening, and before any baseline assessment,
* Has clinically apparent tense effusion of the target knee,
* Has had viscosupplementation in any joint including the target knee within 9 months prior to Screening,
* Has concomitant inflammatory disease or other condition that affects the joints (e.g. rheumatoid arthritis, metabolic bone disease, psoriasis, gout, symptomatic chondrocalcinosis and active infection, etc.,)
* Symptomatic OA of the contralateral knee or of either hip that is not responsive to paracetamol and requires other therapy,
* Has related hypersensitivities to avian proteins and/or any components of hyaluronan-based injection devices,

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (21):
- Belgium (4):
  - Hopital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Gastuisberg Leuven, Leuven
  - CHU Liege, Liège
- Czechia (4):
  - Faculty Hospital Bohunice, Brno
  - Institute of Rheumatology, Prague
  - Faculty Thomayer Hospital, Prague
  - Faculty Hospital Motol, Prague
- France (5):
  - Hopital Henri Mondor, Créteil
  - CHU Dupuytren, Limoges
  - Hopital de la Conception, Marseille
  - Hopital Rangueil, Toulouse
  - CHU Hopital Trousseau, Tours
- Johanna-Etienne Krankenhaus, Neuss, Germany
- Netherlands (2):
  - AMC/UVA, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
- United Kingdom (5):
  - University Hospital of Wales, Cardiff
  - Kings College Hospital, London
  - Trafford General Hospital, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nuffield Orthopaedic Centre, Oxford

REFERENCES:
- [Derived] Chevalier X, Jerosch J, Goupille P, van Dijk N, Luyten FP, Scott DL, Bailleul F, Pavelka K. Single, intra-articular treatment with 6 ml hylan G-F 20 in patients with symptomatic primary osteoarthritis of the knee: a randomised, multicentre, double-blind, placebo controlled trial. Ann Rheum Dis. 2010 Jan;69(1):113-9. doi: 10.1136/ard.2008.094623. PMID 19304567

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 329 participants enrolled and 76 screening failures. One participant was randomised to the Synvisc group but received Saline in error; counted in the Saline group for safety analyses (Safety population) and in the Synvisc group for efficacy analyses (Intent-to-treat population) in both study periods.
Groups:
- Synvisc: Participants with symptomatic primary osteoarthritis (OA) of the knee received a single injection of 6 mL hylan G-F 20 (Synvisc) during the Initial Treatment Period. Participants from both treatment arms had the opportunity to receive an additional 6 mL hylan G-F 20 (Synvisc) during the Repeat Treatment Period.
- Saline Control: Participants (control group) with symptomatic primary osteoarthritis (OA) of the knee received a single injection of 6 mL phosphate buffered saline during the Initial Treatment Period.
Period: Initial Treatment Period
Arm/Group | Synvisc | Saline Control
Started | 123 (Safety population) | 130 (Safety population)
Intent to Treat Population | 124 | 129
Completed | 114 | 118
Not Completed | 9 | 12
Not completed — Adverse Event | 1 | 3
Not completed — Non-compliant | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 6 | 4
Not completed — Other | 0 | 2
Period: Repeat Treatment Period
Arm/Group | Synvisc | Saline Control
Started | 160 (Safety population: 77 Synvisc + 83 Saline Control participants from the Initial Treatment period.) | 0
Completed | 158 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Synvisc: Participants with symptomatic primary osteoarthritis (OA) of the knee received a single injection of 6 mL hylan G-F 20 (Synvisc) during the Initial Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Synvisc | Saline Control | Total
Number analyzed (Participants) | 124 | 129 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.64) | 62.5 (9.17) | 63.0 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 88 | 180
  Male | 32 | 41 | 73
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 118 | 125 | 243
  Black | 5 | 3 | 8
  Hispanic | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Knee Pain Over the Course of the 26-week Initial Treatment Period As Measured by Participants Using the Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale Version 3.1 (WOMAC LK 3.1) A (Pain) Subscale
Description: The change from baseline over the course of the 26-week initial treatment period using participants' assessment of pain. Mean scores were used for baseline (day 0) and for all visits up to week 26 (weeks 4, 8, 12, 18 and 26). The WOMAC Pain Subscale has a score range of 0-4, where 0=no pain and 4=extreme pain.
Time Frame: Day 0, up to week 26
Population: Intent-To-Treat (ITT) population which included all participants randomized to study treatment on Day 0.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Synvisc | Saline Control
Number analyzed (Participants) | 124 | 129
units on a scale | -0.84 (0.060) | -0.69 (0.058)
Statistical Analysis 1: Comparison: Synvisc vs Saline Control; Test type: Superiority or Other; p = 0.047, ANCOVA; The repeated measures ANCOVA model included terms for treatment, site, time and time-by-treatment interaction; the baseline score was a covariate

2. Secondary Outcome: Change From Baseline in Knee Pain at Week 26 As Measured by Participants Using the Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale Version 3.1 (WOMAC LK 3.1) A (Pain) Subscale
Description: The change from baseline to week 26 using participants' assessment of pain. The WOMAC Pain Subscale has a score range of 0-4, where 0=no pain and 4=extreme pain.
Time Frame: Day 0, Week 26
Population: Intent-To-Treat (ITT) population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Synvisc | Saline Control
Number analyzed (Participants) | 124 | 129
units on a scale | -0.76 (0.07) | -0.58 (0.07)
Statistical Analysis 1: Comparison: Synvisc vs Saline Control; Test type: Superiority or Other; p = 0.064, ANCOVA

3. Secondary Outcome: Participants Level of Pain While Walking at Week 26 As Measured by Participants Using the Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale Version 3.1 (WOMAC LK 3.1) A1 (Walking Pain) Subscale
Description: Participants categorized the pain they felt while walking using the WOMAC LK 3.1) A1 (Walking Pain) Subscale. The scale rates pain as none, mild, moderate, severe and extreme.
Time Frame: Week 26
Population: Intent-To-Treat (ITT) population
Measure: Number; unit: participants
Arm/Group | Synvisc | Saline Control
Number analyzed (Participants) | 115 | 117
participants
  None | 17 | 13
  Mild | 45 | 39
  Moderate | 41 | 42
  Severe | 11 | 19
  Extreme | 1 | 4
Statistical Analysis 1: Comparison: Synvisc vs Saline Control; Estimate of Odds Ratio (Placebo/Synvisc-One) using WOMAC A1 data at Week 26; Test type: Superiority or Other; p = 0.022, Generalized Estimating Equations (GEE); Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.35 to 0.92]

4. Secondary Outcome: Change From Baseline Over the Course of the 26-week Initial Treatment Period in Physical Function Measured by Participants Using the Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale (WOMAC LK Version 3.1) C (Function) Subscale
Description: The change from baseline over the course of the 26-week initial treatment period using participants' assessment of physical function. Mean scores were used for baseline (day 0) and for all visits up to week 26 (weeks 4, 8, 12, 18 and 26). The WOMAC Function Subscale has a score range of 0-4 to assess the degree of difficulty completing tasks within the past 48 hours, where 0=no difficulty and 4=extreme difficulty.
Time Frame: Day 0, up to week 26
Population: Intent-To-Treat (ITT) population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Synvisc | Saline Control
Number analyzed (Participants) | 124 | 129
units on a scale | -0.66 (0.061) | -0.63 (0.059)
Statistical Analysis 1: Comparison: Synvisc vs Saline Control; Test type: Superiority or Other; p = 0.679, ANCOVA

5. Secondary Outcome: Change From Baseline at Week 26 in Physical Function Measured by Participants Using the Western Ontario and McMaster Universities Osteoarthritis Index Likert Scale (WOMAC LK Version 3.1) C (Function) Subscale
Description: The change from baseline to week 26 using participants' assessment of physical function. The WOMAC Function Subscale has a score range of 0-4 to assess the degree of difficulty completing tasks within the past 48 hours, where 0=no difficulty and 4=extreme difficulty.
Time Frame: Day 0, Week 26
Population: Intent-To-Treat (ITT) population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Synvisc | Saline Control
Number analyzed (Participants) | 124 | 129
units on a scale | -0.59 (0.076) | -0.48 (0.074)
Statistical Analysis 1: Comparison: Synvisc vs Saline Control; Test type: Superiority or Other; p = 0.266, ANCOVA

6. Secondary Outcome: Participant Global Assessment (PTGA) of the Target Knee Osteoarthritis Condition at Week 26
Description: The Participant Global Assessment (PTGA) was used by participants to rate their osteoarthritis (OA). PTGA uses 5 scoring levels: Very well=0, Well=1, Fair=2, Poor=3, Very poor=4.
Time Frame: Week 26
Population: Intent-To-Treat (ITT) population
Measure: Number; unit: participants
Arm/Group | Synvisc | Saline Control
Number analyzed (Participants) | 115 | 117
participants
  Very Well | 9 | 2
  Well | 33 | 27
  Fair | 50 | 54
  Poor | 21 | 31
  Very Poor | 2 | 3
Statistical Analysis 1: Comparison: Synvisc vs Saline Control; Model-based estimate of Odds Ratio (Placebo/Synvisc-One) using PTGA data at Week 26; Test type: Superiority or Other; p = 0.005, Generalized Estimating Equations (GEE); Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.31 to 0.82]

7. Secondary Outcome: Clinical Observer Global Assessment (COGA) of the Target Knee Osteoarthritis (OA) Condition at Week 26
Description: The Blinded Clinical Observer gave a global assessment (COGA) of the target knee OA. COGA uses 5 scoring levels: Very well=0, Well=1, Fair=2, Poor=3, Very poor=4.
Time Frame: Week 26
Population: Intent-To-Treat (ITT) population
Measure: Number; unit: participants
Arm/Group | Synvisc | Saline Control
Number analyzed (Participants) | 115 | 117
participants
  Very Well | 13 | 8
  Well | 37 | 31
  Fair | 38 | 38
  Poor | 22 | 34
  Very Poor | 5 | 6
Statistical Analysis 1: Comparison: Synvisc vs Saline Control; Model-based estimate of Odds Ratio (Placebo/Synvisc-One) using COGA data at Week 26; Test type: Superiority or Other; p = 0.025, Generalized Estimating Equations (GEE); Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.34 to 0.93]

8. Secondary Outcome: Participants Classified as Responders Per the Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Criteria at Week 26
Description: Participants were classified as a positive responder if at least one of the following two conditions were met:
  1. A significant improvement in either the pain (WOMAC A) or physical function (WOMAC C) subscales, defined as both a ≥ 50% improvement from Baseline and an absolute change from Baseline of ≥ 20 normalised units (NU), OR
  2. Improvement in at least 2 of 3 subscales - pain (WOMAC A), physical function (WOMAC C) or Participant Global Assessment (PTGA). Improvement for all three scales is defined as ≥ 20% improvement from Baseline and an absolute change from Baseline of ≥ 10 NU
Time Frame: Week 26
Population: Intent-To-Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Synvisc | Saline Control
Number analyzed (Participants) | 123 | 129
participants
  Responder - meets OMERACT-OARSI criteria | 73 | 66
  NonResponder -does not meet OMERACT-OARSI criteria | 43 | 52
  NonResponder - Withdrew Before Study Completion | 7 | 11
Statistical Analysis 1: Comparison: Synvisc vs Saline Control; Estimate of Odds Ratio (Placebo/Synvisc-One) using Responder classification data at Week 26; Test type: Superiority or Other; p = 0.156, Generalized Estimating Equations (GEE); Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.41 to 1.16]

ADVERSE EVENTS:
Time Frame: Initial treatment period: Day 1 to Week 26. Repeat treatment period: Week 26 to Week 30.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Events are listed independent of relationship to treatment reported.
Groups:
- Synvisc - Initial Treatment Period: Participants with symptomatic primary osteoarthritis (OA) of the knee received a single injection of 6 mL hylan G-F 20 (Synvisc) during the Initial Treatment Period (up to week 26).
- Saline Control - Initial Treatment Period: Participants (control group) with symptomatic primary osteoarthritis (OA) of the knee received a single injection of 6 mL phosphate buffered saline during the initial treatment period.
- Synvisc - Repeat Treatment Period: Participants from the Synvisc Initial Treatment Period had the opportunity to receive 6 mL hylan G-F 20 (Synvisc) during the Repeat Treatment Period (weeks 26-30).
- Synvisc (From Saline Control) - Repeat Treatment Period: Participants from the Saline Control Initial Treatment Period had the opportunity to receive 6 mL hylan G-F 20 (Synvisc) during the Repeat Treatment Period (weeks 26-30).
Arm/Group | Synvisc - Initial Treatment Period | Saline Control - Initial Treatment Period | Synvisc - Repeat Treatment Period | Synvisc (From Saline Control) - Repeat Treatment Period
Serious Adverse Events (participants affected / at risk) | 5/123 | 3/130 | 0/77 | 2/83
Other Adverse Events (participants affected / at risk) | 70/123 | 77/130 | 9/77 | 11/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synvisc - Initial Treatment Period (N=123) | Saline Control - Initial Treatment Period (N=130) | Synvisc - Repeat Treatment Period (N=77) | Synvisc (From Saline Control) - Repeat Treatment Period (N=83)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synvisc - Initial Treatment Period (N=123) | Saline Control - Initial Treatment Period (N=130) | Synvisc - Repeat Treatment Period (N=77) | Synvisc (From Saline Control) - Repeat Treatment Period (N=83)
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 1 | 1 | 1 | 2
Malaise (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 3 | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0
Dental caries (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0 | 0 | 0
Infected insect bite (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 4 | 7 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Mastitis (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 7 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 1 | 0 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0
Helicobacter pylori identification test positive (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 30 | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 10 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 7 | 7 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 10 | 13 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 | 7 | 0 | 1
Joint warmth (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cervical root pain (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 9 | 15 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 1 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, principal investigator (PI) can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.